CLINICAL TRIAL: NCT01217060
Title: Phase IIB Study of Trimodality Management of Clinical T1bN0M0 Cancers of the Esophagus
Brief Title: Trimodality Management of T1b Esophageal Cancers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-0333; NCI-2012-01902 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2010-10-06; First posted 2010-10-08 (Estimated); Results first posted 2021-04-13 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Esophageal Cancer
Keywords: Adenocarcinoma; Squamous cell carcinoma; Thoracic esophagus; Gastroesophageal junction; Chemoradiotherapy; Esophagectomy; 5-Fluorouracil; Docetaxel; Radiation; Radiotherapy; XRT; IMRT; Taxotere; Adrucil; Efudex; Dexamethasone; Decadron
MeSH Terms: conditions — Esophageal Neoplasms; Adenocarcinoma; Carcinoma, Squamous Cell | interventions — Docetaxel; Fluorouracil; Radiotherapy; Esophagectomy; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Docetaxel + 5-FU + Radiation + Surgery (Experimental): Docetaxel 20 mg/m2 given by vein (IV) once a week up to 5 1/2 weeks. Dexamethasone 10 mg IV 30 minutes prior to weekly Docetaxel. 5-FU 300 mg/m2 IV, continuously for 96 hours 5 days a week for about 5 1/2 weeks. Radiation 50.4 Gy (1.8G/Fx/day) for about 5 1/2 weeks. Surgery to remove part of esophagus and nearby lymph nodes, approximately 8 to 10 weeks after completing chemoradiation.
  Interventions: Drug: Docetaxel; Drug: 5-FU; Radiation: Radiotherapy; Procedure: Esophagectomy; Drug: Dexamethasone

INTERVENTIONS:
Drug: Docetaxel — 20 mg/m2 given by vein (IV) over 1 hour once a week for up to 5 1/2 weeks.
  Other Names: Taxotere
Drug: 5-FU — 300 mg/m2 given by vein, continuously for 96 hours a week for about 5 1/2 weeks.
  Other Names: Adrucil; Efudex; 5-Fluorouracil
Radiation: Radiotherapy — 50.4 Gy (1.8G/Fx/day) for about 5 1/2 weeks, Monday through Friday.
  Other Names: Radiation Therapy
Procedure: Esophagectomy — Surgery to remove part of esophagus and nearby lymph nodes, approximately 8 to 10 weeks after completing chemoradiation.
  Other Names: Surgical Resection
Drug: Dexamethasone — 10 mg IV 30 minutes prior to weekly Docetaxel.
  Other Names: Decadron

SUMMARY:
The goal of this clinical research study is to learn if giving chemotherapy and radiation therapy before surgery for early-stage esophageal cancer can help to control the disease and if so, for how long. The safety of this treatment will also be studied.

DETAILED DESCRIPTION:
The Study Treatment:

5-fluorouracil and docetaxel are designed to stop the growth of cancer cells, which may cause the cells to die. Docetaxel may also damage blood vessels in tumor tissue.

The radiation therapy in this study will be either intensity modulated radiation therapy (IMRT), which is a form of photon-based radiation therapy, or proton beam therapy (PBT). This will be up to your doctor. Both IMRT and PBT are designed to give radiation to the tumor area and limiting radiation exposure to nearby organs such as the lungs, heart, and spinal cord.

The surgery in this study removes part of the esophagus and nearby lymph nodes. The type of surgery will be the doctor's decision based on the location of the tumor in the esophagus. It will either be laparoscopic surgery (a minimally invasive procedure through small holes made in the abdomen) or open surgery (through the chest wall).

Study Treatment Administration:

If you are found to be eligible to take part in this study, you will receive radiation therapy and chemotherapy on the following schedule for up to 5 1/2 weeks. If there are holidays on the scheduled treatment days, the schedule may be slightly different and the study staff will discuss this with you.

* Radiation therapy will be given Monday through Friday. This will take about 30 minutes, including about 10-15 minutes for the radiation treatment.
* 5-fluorouracil will be given by vein, continuously for about 96 hours a week (Monday through Friday).
* Docetaxel will be given by vein over about 1 hour, 1 time a week (on Mondays).

  5-fluorouracil will be given using a portable pump about the size of a personal CD player. You will need to carry this portable pump with you for about 96 hours each week.

Docetaxel will be given through a central venous catheter. A central venous catheter is a sterile flexible tube that will be placed into a large vein while you are under local anesthesia. Your doctor will explain this procedure to you in more detail, and you will be required to sign a separate consent form for this procedure. The catheter will be removed at the end of Week 5.

Before every dose of docetaxel, you will receive dexamethasone to lower the risk of side effects. Dexamethasone will be given by vein over a few seconds.

Your doctor will let you know if and when you are eligible to have surgery. In this study, the surgery must be performed within 8-10 weeks after you finish chemotherapy and radiation therapy. You will be asked to sign a separate consent form that describes the surgery and anesthesia (numbing medicine) and their risks in more detail. The screening tests that will help your doctor decide if you are eligible to have surgery include the scans and endoscopy described below (4-6 weeks after radiation and chemotherapy).

You will no longer be able to receive radiation and chemotherapy if the disease gets worse or intolerable side effects occur. You will not be able to have surgery if the doctor decides surgery is not in your best interest (for example, if the disease or your general health gets worse).

Study Visits:

During Study Therapy:

Blood (about 3 tablespoons) will be drawn for routine tests during Week 3 of radiation and chemotherapy.

Follow-Up:

At 4-6 weeks after your last dose of radiation and chemotherapy, the following tests and procedures will be performed:

* You will have a CT scan of the chest and a whole-body PET/CT scan to check the status of the disease.
* You may have an endoscopy of your esophagus with 1 or more biopsies of the tumor to check the status of the disease. The number of biopsies you have will be the doctor's decision at the time of the procedure, based on the status and location of the disease.
* Blood (about 3 tablespoons) will be drawn for routine tests.
* You will fill out 3 quality-of-life questionnaires. This should take about 10-15 minutes.

About 4 weeks after surgery, you will fill out 3 quality-of-life questionnaires. You will then fill out 2 quality-of-life questionnaires at 6 of your routine follow-up visits after surgery.

Every 3-6 months in the first 3 years after your last dose of radiation and chemotherapy, then every 6 months in the next 2 years, and every year after that from then on, the following tests and procedures will be performed:

* You will have a CT scan of the chest or a whole-body PET/CT scan to check the status of the disease.
* You will have an endoscopy of your esophagus to check the status of the disease during every follow-up visit in Year 1. After that, you will have an endoscopy of your esophagus at follow-up visits anytime the doctor decides it is needed. You will have 1 or more tumor biopsies at these follow-up visits if the doctor decides they are needed, based on the status and location of the disease. This will be decided at the time of the endoscopy.

Biomarker Testing:

If leftover tumor tissue is available from before you joined the study, the leftover tissue will be used for genetic biomarker testing. If you do not have leftover tumor tissue available from before you joined the study, leftover tissue from study procedures will be used for genetic biomarker testing.

This is an investigational study. Docetaxel and 5-fluorouracil are FDA approved and commercially available to treat esophageal cancer. However, it is investigational to give these drugs to patients with early-stage esophageal cancer.

It is investigational to give the combination of chemotherapy, radiation therapy, and surgery to patients with early-stage esophageal cancer.

Up to 30 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically documented adenocarcinoma or squamous cell carcinoma of the thoracic esophagus or gastroesophageal junction that are staged as T1b using endoscopic ultrasound (EUS) or from a large biopsy (either criteria # 1 or #2 can be met for eligibility).
2. Patients who undergo a diagnostic Endoscopic Mucosal Resection (EMR) and have a diagnosis of T1b stage established.
3. Performance score Karnofsky Performance Scale (KPS) 80-100.
4. Patients should be surgical candidates for esophagectomy and should have no contraindications for chemotherapy or radiation.
5. Negative pregnancy test for women of child bearing potential. They must agree to adequate contraception.
6. Complete blood count (CBC) and complete metabolic panel (chemo-14: Glucose, Calcium, Albumin, Total Protein, Sodium, Potassium, CO2, Chloride, Blood Urea Nitrogen (BUN), Creatinine, Alkaline Phosphatase, ALT (SGPT), AST (SGOT), and Bilirubin) to assess adequate hematologic, renal and hepatic functioning will be obtained. The values are as follows: Adequate hematologic (White Blood Count (WBC) >2,500/uL, platelets > 75,000/uL), renal (creatinine clearance > 50 mL/min), and liver function (bilirubin <=1.5 fold the upper limit of normal and liver enzymes < 3 fold the upper limit of normal).
7. Based on the risk factors and propensity of lymph node metastasis (LNM) and poorer survivals seen in retrospective studies as discussed in the introduction, only patients with any one (1) of high risk features such as LVI, tumors >1.2 cm, and high grade will be enrolled (Grade is the pathologic term defining the degree of differentiation. Grade 1 is well differentiated, Grade 2 is moderately differentiated, and Grade 3 is poorly differentiated).

Exclusion Criteria:

1. Prior radiation to the chest
2. Previous or concomitant cancers other than 1) curatively treated carcinoma in situ of cervix, basal cell of the skin, curative treatment for transitional cell carcinoma of the bladder, and early stage cancers at another non-overlapping site that was treated more than 3 years ago for cure.
3. Pregnant or breast-feeding females
4. Clinically significant uncontrolled major cardiac, respiratory, renal, hepatic, gastrointestinal or hematologic disease but not limited to: a) active uncontrolled infection b) Symptomatic congestive heart failure, unstable angina, or cardiac dysrrhythmia not controlled by pacer device c) no myocardial infarction within 3 months of registration
5. Known hypersensitivity to docetaxel, 5-fluorouracil, polysorbate-80, or any component of the formulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2010-10 (Actual); Primary Completion 2020-06-14 (Actual); Study Completion 2020-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven H. Lin, MD, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 4 patients were consented to this study, but 1 patient want to get PROTONS treatment instead of IMRT and withdrew consent. 3 patients was treated under this protocol.
Period: Overall Study
Arm/Group | Docetaxel + 5-FU + Radiation + Surgery
Started | 4
Completed | 3
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: 3 out of 4 patients was were consented and treated under this protocol. 1 patients withdrew consent prior to protocol treatment.
Arm/Group | Docetaxel + 5-FU + Radiation + Surgery
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 2
Age, Continuous [Median (Full Range); unit: years] | 67 [56 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3
Karnofsky performance score (KPS) [Count of Participants; unit: Participants] — The Karnofsky Performance Status scores range from 0 to 100. The higher KPS scores, the better treatment outcome. KPS 80 Normal activity with effort; some signs or symptoms of disease. KPS 70 Cares for self; unable to carry on normal activity or to do active work.
  Participants
    KPS≥ 80 | 3
    KPS≥ 70 | 0
Smoking [Count of Participants; unit: Participants]
  Never | 0
  Prior | 3
  Current | 0
Tumor Location [Count of Participants; unit: Participants]
  Cardioesophageal Junction (GEJ) | 2
  Lower (distal) esophgus & GEJ | 1
Tumor Histology- Adenocarcinoma [Count of Participants; unit: Participants] | 3
Moderate to Poorly Differentiation [Count of Participants; unit: Participants] | 3

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Complete Response (PCR) Rate
Description: The primary endpoint for this protocol is to assess the efficacy (pathologic complete response) and safety of Trimodality management (chemoradiotherapy followed by esophagectomy) in patients with clinically staged T1bN0M0 cancer of the esophagus or gastroesophageal junction. This is a single-arm phase IIB trial of chemo-radiation followed by surgery for patients with early stage grade T1b esophageal cancer. The rates of pathologic CR will be tabulated and their possible relationships to baseline covariates assessed by logistic regression. Unadjusted progression free survival time will be estimated by the method of Kaplan and Meier and its possible relationship to baseline covariates assessed by survival regression modeling.
Time Frame: Pathologic Complete Response (PCR) will repeat EGD with biopsy to assess for clinical response to therapy after chemoradiation four to six weeks.
Population: There are no statistical data analysis results available due to the protocol terminated early due to low rate of accrual, changes in treatment paradigm (patients are going for local excision for T1b esophageal cancer). We incorporated the analysis of those patient to the paper of a retrospective cohort, since the 4 patients themselves were not reportable.
Arm/Group | Docetaxel + 5-FU + Radiation + Surgery
Number analyzed (Participants) | 0

2. Secondary Outcome: Disease-free Survival (DFS) Time
Description: Disease-free survival (DFS) defined as the time to disease progression or death. DFS calculated from the time of surgery to disease progression or death. Followed for disease recurrence every 3-6 months in the first 3 years after last dose of radiation and chemotherapy, then every 6 months in the next 2 years, then every year.
Time Frame: Time to disease progression or death, up to 6 years
Population: There are no statistical data analysis results available because this protocol termination early due to low rate of accrual, changes in treatment paradigm (patients are going for local excision for T1b esophageal cancer).
Arm/Group | Docetaxel + 5-FU + Radiation + Surgery
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From date of protocol registration until the date of documented development of adverse events (AEs) , assessed at the end of the 30-day period following surgery
Description: Toxicity was documented according to the Common Terminology Criteria for Adverse Events (CTCAE) V4.0 during the 10-week period beginning at the start of chemo-radiation and ending at the time of surgery, and post-surgery mortality (PostDeath), defined as death due to any cause during the 30-day period following surgery.
Arm/Group | Docetaxel + 5-FU + Radiation + Surgery
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 3/3
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Docetaxel + 5-FU + Radiation + Surgery (N=3)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Diaphoresis (Metabolism and nutrition disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Dysgeusia (Nervous system disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 3 (4)
Esophagitis (Gastrointestinal disorders) | 2 (2)
Fatigue (General disorders) | 3 (5)
Lymphopenia (Investigations) | 1 (1)
Mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Neuropathy (Nervous system disorders) | 1 (1)
Odynophagia (Gastrointestinal disorders) | 3 (3)
Radiation Dermatitis (Skin and subcutaneous tissue disorders) | 1 (2)
Rash (Hand-Foot skin reaction) (Skin and subcutaneous tissue disorders) | 1 (2)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Weight loss (Investigations) | 1 (1)

LIMITATIONS AND CAVEATS:
There are no statistical data analysis results available due to the protocol terminated early due to low rate of accrual, changes in treatment paradigm (patients are going for local excision for T1b esophageal cancer). We incorporated the analysis of those patient to the paper of a retrospective cohort, since the 4 patients themselves were not reportable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-12): https://cdn.clinicaltrials.gov/large-docs/60/NCT01217060/Prot_SAP_000.pdf